CLINICAL TRIAL: NCT00000221
Title: Alternate-Day Buprenorphine Administration. Phase I
Brief Title: Alternate-Day Buprenorphine Administration. Phase I - 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-06969-3; R01-06969-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-11

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to determine if two times a subject's daily maintenance dose will hold for 48 hours without changes in agonist and antagonist effects.

ELIGIBILITY:
Please contact site for information.

Ages: 28 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1992-04

PRIMARY OUTCOMES:
Drug use
Opioid withdrawal
Opioid agonist effects
Dose identification
Pupil diameter

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States

REFERENCES:
- [Background] Amass L, Bickel WK, Higgins ST, Badger GJ. Alternate-day dosing during buprenorphine treatment of opioid dependence. Life Sci. 1994;54(17):1215-28. doi: 10.1016/0024-3205(94)00848-5. PMID 8164503